CLINICAL TRIAL: NCT02788253
Title: Comparison of the Mallampati Classification and Best Visible Mallampati for Prediction of Difficult Tracheal Intubation
Brief Title: Mallampati Classification vs Best Visible Mallampati for Prediction of Difficult Tracheal Intubation
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: A15-D11-VOL.24
Record Dates: First submitted 2016-02-09; First posted 2016-06-02 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2017-03

CONDITIONS: Intubation; Difficult
Keywords: Mallampati; Intubation difficult; Mask ventilation difficult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Mallampati score (classification of the visibility of oropharyngeal structures) should be performed in the sitting position, head in the neutral position, mouth widely open, and tongue protrudes, without phonation. However, phonation, and position modify the visibility of oropharyngeal structures and thus the Mallampati score.

We aimed at evaluating the predictive value of the best observable Mallampati score as compare to the recommended Mallampati score.

DETAILED DESCRIPTION:
Mallampati score (classification of the visibility of oropharyngeal structures) should be performed in the sitting position, head in the neutral position, mouth widely open, and tongue protrudes, without phonation. However, phonation, and position modify the visibility of oropharyngeal structures and thus the Mallampati score.

We aimed at evaluating the predictive value of the best observable Mallampati score as compare to the recommended Mallampati score.

This is a single center prospective observational study comparing the original Mallampati classification to the best visible Mallampati classification.

Data and variables concerning airway management during induction of general anesthesia are recorded on a specific record sheet.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled or unscheduled surgery
* Airway evaluation possible in both sitting and supine position

Exclusion Criteria:

* surgery of the neck, face, and upper airway
* lung and thoracic surgery
* pregnancy
* orotracheal intubation not indicated during surgery
* nasotracheal intubation required for surgery
* selective intubation required for surgery
* emergency surgery and procedure

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients (16 years older) scheduled for vascular, orthopedic, urologic, gynecologic, and abdominal surgery.
  Airway evaluation must be possible in full Orotracheal intubation required for general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 3244 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with difficult airway management | 1 day
  Occurence of either difficult tracheal intubation or difficult face mask ventilation or both
  Difficult tracheal intubation was defined as an orotracheal intubation requiring more than 2 laryngoscopies, or lasting more than 10 min, or requiring an alternate device (gum elastic bougie, supraglottic device, videolaryngoscope) Difficult mask ventilation was defined as the inability for the anesthesiologist to provide adequate ventilation because of one or more of the following problems: inability for the unassisted anesthesiologists to maintain oxygen saturation > 92% using 100% oxygen, excessive gas leak requiring use of the oxygen flush valve more than twice, excessive insufflation pressure (> 25 cmH2O), absence of spirometric measures of exhaled gas flow or a tidal volume < 3ml/kg, absence or inadequate exhaled carbon dioxide, necessity to perform two-handed mask ventilation

SECONDARY OUTCOMES:
Number of patient with difficult Face Mask Ventilation | 1 day
  Difficult mask ventilation was defined as the inability for the anesthesiologist to provide adequate ventilation because of one or more of the following problems: inability for the unassisted anesthesiologists to maintain oxygen saturation > 92% using 100% oxygen, excessive gas leak requiring use of the oxygen flush valve more than twice, excessive insufflation pressure (> 25 cmH2O), absence of spirometric measures of exhaled gas flow or a tidal volume < 3ml/kg, absence or inadequate exhaled carbon dioxide, necessity to perform two-handed mask ventilation
Number of patients with difficult tracheal intubation | 1 day
  Difficult tracheal intubation was defined as an orotracheal intubation requiring more than 2 laryngoscopies, or lasting more than 10 min, or requiring an alternate device (gum elastic bougie, supraglottic device, videolaryngoscope)

OTHER OUTCOMES:
Correct Reclassification rate of patients by best view of Mallampati | 1 day
  Statistical analysis using reclassification methods (net reclassification improvement)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Hanouz, M.D.,Ph.D., Principal Investigator — University Hospital, Caen
Locations (1):
- University Hospital of Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanouz JL, Lefrancois V, Boutros M, Fiant AL, Simonet T, Buleon C. Comparison of the modified Mallampati classification score versus the best visible Mallampati score in the prediction of difficult tracheal intubation: a single-centre prospective observational study. Can J Anaesth. 2024 Oct;71(10):1353-1362. doi: 10.1007/s12630-024-02815-0. Epub 2024 Aug 15. PMID 39147992